CLINICAL TRIAL: NCT01469455
Title: An Open Label, Non-randomized, First-in-human, Multi-centre Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Locally Administered DT01 in Combination With Radiotherapy and Concomitant Dose of Chloroquine in Patients With Local Metastatic Melanoma With Relapsed Cutaneous/Subcutaneous Tumors Including Melanoma-in-transit
Brief Title: DNA Repair Inhibitor & Irradiation on Melanoma
Acronym: DRIIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DNA Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DT01-01
Record Dates: First submitted 2011-10-24; First posted 2011-11-10 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Local Metastatic Melanoma
Keywords: Local metastatic melanoma; relapsed cutaneous/subcutaneous tumors; melanoma-in-transit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DT01 (Experimental)
  Interventions: Drug: DT01

INTERVENTIONS:
Drug: DT01 — DT01 starting dose will be 16 mg and it is planned to be increased to 32, 48 mg and 64 mg, or higher.
  DT01 will be administered 3 times a week (e.g., Mondays, Wednesdays and Fridays) over 2 weeks (6 administrations of DT01 in total) at least 3 hours prior to the radiotherapy sessions.

SUMMARY:
Phase I trial will be conducted in patients suffering local metastatic melanoma with relapsed cutaneous/subcutaneous tumors including melanoma-in-transit. Based on the preclinical data package, DNA Therapeutics has considered that the risk-benefit ratio of DT01 supports the initiation of a phase I clinical study in this population. The recommended starting dose of DT01 for the first injection to human was based on NOAELs and Maximum Recommended Starting Dose (MRSD) calculations and by considering both local and systemic approaches. It was set at 16 mg (4 mg per injection site, 2 injections per tumor, 2 tumors to be treated). This starting dose will be increased up to 96 mg if no DLT occurred during dose escalation.

DT01 will be locally administered by peritumoral subcutaneous and/or intratumoral injections in combination with hypo-fractionated radiotherapy (RT) (10x 3 Gy) and chloroquine (100 mg oral QD) starting one week before DT01 and RT treatments. DT01 will be administered 3 times a week during two weeks; The study will be an open, non-randomised, multicentre, phase I dose escalation (16, 32, 48, 64 and 96 mg) safety study with a 3+3 design.

The purpose of this study will be to evaluate the safety, tolerance, pharmacokinetics of DT01 in association with palliative radiotherapy and to evaluate pharmacodynamics and the anti-tumor activity of DT01 according to RECIST criteria on day 26, 40 and 54. The duration of response (Time-To-Local Recurrence, TTLR), will be monitored 3, 6, 9 and 12 months after the beginning of the DT01 treatment.

DETAILED DESCRIPTION:
According to the WHO, the incidence of melanoma is 199,627 worldwide in 2008, of which the melanoma-in-transit is about 4%. When melanoma spreads, it does so by the lymphatic system which drains to the regional lymph nodes. Uncommonly, melanoma can become trapped in the lymphatic vessels and grow to cause tumor nodules in the skin and subcutaneous tissues between the primary site and the regional lymph node basin. These nodules are termed in-transit metastases and carry an ominous prognosis. The American Joint Committee on Cancer (AJCC) defines such in-transit metastases as any skin or subcutaneous metastases that are more than 2 cm from the primary lesion but are not beyond the regional nodal basin. The 2010 tumor node metastasis (TNM) staging system considers the melanoma-in-transit a N2c stage when they arise in the absence of nodal metastases.

The current treatment options (approved or in late stage development) are:

* Local excision, if there are only a few;
* Isolated limb perfusion (local high dose chemotherapy);
* Systemic chemotherapy (Dacarbazine, Temozolomide, Cis-platine);
* Targeted therapy (B-raf inhibitors: Vemurafenib and Dabrafenib; MEK inhibitor: Trametinib);
* Immunotherapy (Ipilimumab, Nivolumab, Pembrolizumab, OncoVEX GM-CSF, Tumor Infiltrating Lymphocytes and interleukin-2 [IL-2]);
* Radiotherapy;
* Photodynamic therapy;
* Laser vaporization. With rare exceptions, none of these treatments are curative. Immunotherapy results in prolongation of survival although overall response rate remains low (ref: oncovex phase II study).

According to the Sponsor's clinical development strategy and plan, the local metastatic melanoma with relapsed cutaneous/subcutaneous tumors, including melanoma-in-transit, has been chosen as the 1st indication for evaluating safety, tolerance and PK of DT01 in combination with a palliative radiotherapy (10x3 Gy). The presence of multiple cutaneous/subcutaneous tumor should provide an initial clinical evaluation of the safety and skin tolerance of the combined treatment of DT01 and 10x3 Gy irradiation, as well as a preliminary assessment of anti-tumor activity (proof of concept) of DT01 to sensitize and improve the response rate of radiotherapy (estimated about 50% response rate), and to delay local relapse.

Based on the pharmacologically active dose in human melanoma xenografted tumor in mice and the wide safety margin estimated from the toxicology data, the starting dose of 16 mg and the planned dose escalation represent a conservative approach for titration. The dose escalation will provide valuable information about the safety, tolerance and preliminary efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic melanoma with relapsed cutaneous tumors, including melanoma-in-transit, who are not eligible for immediate surgery or refractory to conventional treatment;
* Patients with at least two measurable tumors of ≤ 4cm in largest diameter. Treated tumors must not be previously irradiated.

The consideration of tumor size and number for the 5th and expansion cohorts can be revised based on the observation for the 4 first cohorts, in particular the initial indication of efficacy, after an agreement between Principal Investigators, the DSMB and the Sponsor.

* Normal haematopoietic function as assessed by a complete blood count including differential count.

  i.Absolute neutrophil count ≥ 1.5 x 109/L; ii.Platelet count ≥ 100 x 109/L; iii.Haemoglobin ≥ 10 g/dL (transfusions are permitted);
* No clinically relevant abnormalities in the results of the pre-study laboratory tests:

  i.Creatinine ≤ 1.5 times UNL (upper normal of the limit) ; ii.Bilirubin ≤ 1.5 times UNL; iii.ASAT (SGOT) ≤ 2.5 times the upper limit of normal if no liver metastasis and ≤ 5 times the upper limit of normal in the presence of liver metastasis ; iv.ALAT (SGPT) ≤ 2.5 times the upper limit of normal if no liver metastasis and ≤ 5 times the upper limit of normal in the presence of liver metastasis;
* Age ≥18 years old;
* The patient is willing and able to comply with the protocol for the duration of the study, including 1 day of hospitalization for PK sample at Day 1 and scheduled follow-up visits and examinations to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Exclusion Criteria:

* Presence of any serious concomitant systemic disorders incompatible with the study (e.g. active infection);
* Known or suspected Central Nervous System (CNS) metastases including leptomeningeal metastases (unless the patient has been previously treated and the patient meets the three following criteria: is asymptomatic, has no evidence of active CNS metastases for more than 3 months prior to enrollment, and has no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days);
* Patients with a history of porphyria;
* Patients with active psoriasis;
* Clinically significant hepatic disease (particularly cirrhosis) or renal disease;
* Severe gastrointestinal, neurological and blood disorders;
* Patients receiving anti-vitamin K therapy within 10 days prior to first dose of study treatment (Low Molecular Weight Heparin (LMWH) therapy is allowed);
* Anticancer therapy (chemotherapy, hormone therapy or immunotherapy) within 4 weeks prior to first dose of study treatment and immunotherapy with Ipilimumab, within 3 months prior to first dose of study treatment ;
* Patients receiving cyclosporin within 10 days prior to first dose of study treatment;
* Patients intended to receive any systemic anticancer therapy within 26 days (±2 days) from the anticipated date of the first administration of DT01
* Pregnant or breast-feeding women, or women of child-bearing potential unless effective methods of contraception are used. Child-bearing potential is defined as:

  i.Has experienced menarche, and ii.Has not undergone successful surgical sterilisation, and iii.Is not post-menopausal (amenorrhea > 12 consecutive months or is on Hormone Replacement Therapy (HRT) with a documented plasma or serum FSH > 35 IU/L. iv.Women using oral, implanted, injectable, mechanical or barrier products for the prevention of pregnancy, or who are practising abstinence, or where the partner is sterile (for example, a vasectomy) should be considered to be of child-bearing potential
* Concomitant participation to another study;
* Hypersensitivity to 4-aminoquinoline compounds (chloroquine) or to any of its derivatives;
* HIV and Hepatitis B or C positive patients;
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2
* Retinal or visual field changes attributable to previous chloroquine administration or any other etiology;
* Any reason why, in the Investigator's opinion, the patient should not participate in the study.
* Disease burden judged high, and therefore the patient can not likely benefit from the proposed treatment.
* Significant coagulation abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety analysis, according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4 (NCI-CTCAE v4.0) criteria. | over a period of 54 days
  Tolerability and safety analysis, according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4 (NCI-CTCAE v4.0) criteria.

SECONDARY OUTCOMES:
Profile of pharmacokinetics(PK) | pre-dose,1, 2.5, 4.5, 6.5, 9,24h post dose on Day 1, and pre-dose,4.5h post dose on Day 12
  * Cmax The plasma peak concentration
  * tmax The time to reach the peak concentration
  * AUCt The area under the concentration-time curve from time zero to the last sample with the quantifiable concentration
  * AUC∞ The area under the concentration-time curve from time zero to infinity
  * t½ The terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LE TOURNEAU, MD, Principal Investigator — Institut Curie - National Coordinator; Marie-Françoise AVRIL, MD, Principal Investigator — Groupe Hospitalier Cochin - Hôtel Dieu-Broca; Philippe SAIAG, MD, Principal Investigator — Hospital Ambroise Paré Paris; Céleste LEBBE, MD, Principal Investigator — Hôpital Saint-Louis; Jean-Jacques GROB, MD, Principal Investigator — Hôpital de la Timone; Brigitte DRENO, MD, Principal Investigator — Hôpital hôtel-Dieu; Caroline DUTRIAUX, MD, Principal Investigator — Hôpital Saint-André; Laurent MORTIER, MD, Principal Investigator — Hôpital Claude-Huriez; Eve MAUBEC, MD, Principal Investigator — APHP Hôpital Bichat - Claude Bernard; Luc THOMAS, MD, Principal Investigator — Centre Hospitalier Lyon Sud; Jean-Philippe LACOUR, MD, Principal Investigator — CHU de Nice - Archet 2; Pascal JOLY, MD, Principal Investigator — Hôpital Charles Nicolle
Locations (12):
- France (12):
  - Hôpital Saint-André, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Centre Oscar Lambret, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital hôtel-Dieu, Nantes
  - CHU de Nice - Archet 2, Nice
  - Groupe Hospitalier Cochin - Hôtel Dieu-Broca, Paris
  - Institut Curie, Paris
  - Hôpital Saint-Louis, Paris
  - APHP Hôpital Bichat - Claude Bernard, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Charles Nicolle, Rouen